CLINICAL TRIAL: NCT05370495
Title: A Phase 2, Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Dose-Response, Parallel-Group Study of SY-201 Ophthalmic Solution Versus Vehicle Control in Subjects With Dry Eye Disease
Brief Title: Study of SY-201 Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seinda Pharmaceutical Guangzhou Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY201-CS201
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-masked, parallel, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SY-201 Ophthalmic Solution 2.0% (Experimental): SY-201 Ophthalmic Solution 2.0%
  Interventions: Drug: SY-201 Ophthalmic Solution 2.0%
- SY-201 Ophthalmic Solution 1.0% (Experimental): SY-201 Ophthalmic Solution 1.0%
  Interventions: Drug: SY-201 Ophthalmic Solution 1.0%
- SY-201 Ophthalmic Solution 0.5% (Experimental): SY-201 Ophthalmic Solution 0.5%
  Interventions: Drug: SY-201 Ophthalmic Solution 0.5%
- SY-201 Ophthalmic Solution Vehicle (Placebo Comparator): SY-201 Ophthalmic Solution Vehicle
  Interventions: Drug: SY-201 Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: SY-201 Ophthalmic Solution 2.0% — SY-201 Ophthalmic Solution 2.0%
  Arms: SY-201 Ophthalmic Solution 2.0%
Drug: SY-201 Ophthalmic Solution 1.0% — SY-201 Ophthalmic Solution 1.0%
  Arms: SY-201 Ophthalmic Solution 1.0%
Drug: SY-201 Ophthalmic Solution 0.5% — SY-201 Ophthalmic Solution 0.5%
  Arms: SY-201 Ophthalmic Solution 0.5%
Drug: SY-201 Ophthalmic Solution Vehicle — SY-201 Ophthalmic Solution Vehicle
  Arms: SY-201 Ophthalmic Solution Vehicle

SUMMARY:
This is a phase 2, multi-center, double-masked, randomized, vehicle-controlled, dose-response, parallel-group study designed to evaluate the safety and tolerability and ocular efficacy of SY-201 Ophthalmic Solution versus vehicle over a 60-day treatment period in subjects with dry eye disease (DED).

ELIGIBILITY:
* Inclusion Criteria

  1. Provide written informed consent prior to any study-related procedures.
  2. Are 18 years of age or older.
  3. Are willing and able to follow instructions and can be present for the required study visits for the duration of the study.
  4. Have a Best Corrected Visual Acuity (BCVA) in each eye, using corrective lenses if necessary, of +0.7 logarithm of the minimum angle of resolution (LogMAR) or better as assessed by the Early Treatment of Diabetic Retinopathy Study (ETDRS) at Visit 1.

Exclusion Criteria:

1. Unanesthetized Schirmer test score in either eye <2 mm/5 minutes at Visit 1.
2. Any concomitant treatment or prior ocular procedure or surgery in either eye or alteration of the dose of systemic medications at the time of entry into the study that could interfere in the assessment of the trial
3. Have corneal erosive disease (e.g., confluent staining [National Eye Institute (NEI) grade 4], confluent filaments) or other conditions suggestive of extensive damage of the cornea in either eye.
4. Have a history of glaucoma or intraocular pressure (IOP) >25 mmHg at Visit 1 or a history of elevated IOP (>25 mmHg) in either eye.
5. Wear contact lenses for 14 days prior to Visit 1 or throughout the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lexitas, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Study Eye
Period: Overall Study
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
Started (Randomized) | 50; 50 Study Eye | 51; 51 Study Eye | 51; 51 Study Eye | 49; 49 Study Eye
Withdraw Before Treatment | 1; 1 Study Eye | 0; 0 Study Eye | 1; 1 Study Eye | 1; 1 Study Eye
Received Investigational Product Treatment | 49; 49 Study Eye | 51; 51 Study Eye | 50; 50 Study Eye | 48; 48 Study Eye
Discontinued | 1; 1 Study Eye | 0; 0 Study Eye | 0; 0 Study Eye | 2; 2 Study Eye
Completed | 48; 48 Study Eye | 51; 51 Study Eye | 50; 50 Study Eye | 46; 46 Study Eye
Not Completed | 2; 2 Study Eye | 0; 0 Study Eye | 1; 1 Study Eye | 3; 3 Study Eye

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 50 | 51 | 51 | 49 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 25 | 20 | 86
  >=65 years | 29 | 31 | 26 | 29 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.2) | 64.8 (10.8) | 65.0 (9.2) | 64.2 (13.1) | 64.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 44 | 35 | 155
  Male | 14 | 11 | 7 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 4 | 12
  Not Hispanic or Latino | 47 | 48 | 49 | 45 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 13 | 11 | 10 | 44
  White | 38 | 34 | 40 | 35 | 147
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 51 | 49 | 201

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Corneal Fluorescein Staining (tCFS) at Day 60
Description: Cornea is divided into 5 regions and each region is stained and graded from 0 - 4 (modified National Eye Institute scale (0 (none) to 4 (severe)). Total corneal fluorescein staining score is the sum of the scores from 5 regions (0 -20).
Time Frame: 60 days
Population: Analysis population here is the Per Protocol (PP) Analysis Set (PPAS). PPAS included all subjects who completed study-required treatment and who followed the protocol without significant deviations.
Measure: Mean (Standard Deviation); unit: tCFS score on a scale of 0 - 20
Units Other Than Participants: Study Eyes
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 47 | 48 | 49 | 45
Number analyzed (Study Eyes) | 47 | 48 | 49 | 45
tCFS score on a scale of 0 - 20 | -2.04 (1.989) | -1.65 (2.642) | -2.15 (2.409) | -1.54 (2.598)

2. Primary Outcome: Change From Baseline in Eye Dryness Score (Visual Analog Scale) at Day 60
Description: Eye dryness score as measure by visual analog scale (0 (none) to 100 (severe)) was used to as efficacy meaure for dry eye symptom improvement. This outcome measure focused on self reported extent of eye dryness.
Time Frame: 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on visual analog scale (0 -100)
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 47 | 48 | 49 | 45
Score on visual analog scale (0 -100) | -18.9 (23.3) | -16.9 (19.75) | -20.0 (21.56) | -14.7 (21.56)

3. Secondary Outcome: Change From Baseline in Central Corneal Fluorescein Staining (cCFS) at Day 60
Description: Cornea is divided into 5 regions. The central region is graded from 0 - 4 (modified National Eye Institute scale (0 (none) to 4 (severe)).
Time Frame: 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale of cCFS (mNEI: 0 - 4)
Units Other Than Participants: Study Eyes
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 47 | 48 | 49 | 45
Number analyzed (Study Eyes) | 47 | 48 | 49 | 45
Score on a scale of cCFS (mNEI: 0 - 4) | -0.33 (0.653) | -0.36 (0.933) | -0.44 (0.517) | -0.18 (0.641)

4. Secondary Outcome: Change From Baseline in Symptom Severity Score (Subscale) at Day 60
Description: Symptom severity score sub scale is measured of severity scale of symptoms associated with dry eye using visual analog scale (0 (none) -100 (severe)). This self reported Dry eye symptoms severity score sub scale measures the extent of any ocular discomfort (symptoms), including but not limited to dryness, ocular pain or other type of symptoms.
Time Frame: 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 47 | 48 | 49 | 45
units on a scale 0-100 | -19.8 (23.05) | -19.7 (25.48) | -19.4 (21.09) | -11.5 (19.47)

ADVERSE EVENTS:
Time Frame: 60 days
Description: Complies with clinicaltrials.gov definitions
Arm/Group | SY-201 Ophthalmic Solution 2.0% | SY-201 Ophthalmic Solution 1.0% | SY-201 Ophthalmic Solution 0.5% | SY-201 Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 8/49 | 3/51 | 4/50 | 4/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SY-201 Ophthalmic Solution 2.0% (N=49) | SY-201 Ophthalmic Solution 1.0% (N=51) | SY-201 Ophthalmic Solution 0.5% (N=50) | SY-201 Ophthalmic Solution Vehicle (N=48)
Eye Disorders (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Instillation site irritation (General disorders) | 5 (5) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Collaborative and collegial interaction on presentations and publications.

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT05370495/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT05370495/SAP_001.pdf